CLINICAL TRIAL: NCT05579405
Title: Soluble C-type Lectin-Like Receptor 2 in Stroke Study
Brief Title: sCLEC-2 in Stroke Study
Acronym: CLECSTRO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Yamanashi (Other)
Responsible Party: Principal Investigator, Katsue Suzuki-Inoue M.D. Ph.D., Professor of Department of Clinical and Laboratory Medicine, University of Yamanashi
Other Study IDs: CLEC-0001-02; CS0011 (Other: University of Yamanashi); UMIN000048954 (Other: UMIN-CTR)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Acute Ischemic Stroke; Transient Ischemic Attack
Keywords: Platelet Activation; Soluble C-Type Lectin-Like Receptor 2
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Acute Ischemic Stroke: Ischemic stroke within 24 hours of onset and modified Rankin Scale 0 to 2
- Transient ischemic attack: Transient ischemic attack without MRI positivity within 7 days of onset
- Patient Control: Contemporary patients with neurological symptoms required for differentiation from ischemic stroke or transient ischemic attack

SUMMARY:
Any platelet function tests have not been widely used in the clinical practice of acute cerebrovascular disease because of the concerns in repeatability, economic performance, and simplicity. Soluble C-type lectin-like receptor 2 (sCLEC-2) is a new marker for platelet activation, which can be easily measured by usual blood collection in routine clinical practice. We planned the sCLEC-2 in Stroke (CLECSTRO), which is a prospective cohort study in patients with acute ischemic stroke (AIS) and transient ischemic attack (TIA). We planned the sCLEC-2 in Stroke (CLECSTRO), which is a prospective cohort study in patients with acute ischemic stroke (AIS) and transient ischemic attack (TIA).

The purpose of this study is to evaluate the clinical utility of sCLEC-2 as a biomarker for pathophysiology, differential diagnosis, prediction of prognosis, and monitoring of antiplatelet therapy in patients with AIS and TIA. Subjects are patients with AIS or TIA and control patients required for differentiation from AIS or TIA. The target population is 600 including the patients and the controls. The outcomes include difference in plasma sCLEC-2 level between patients with AIS or TIA and patient controls, correlation between sCLEC-2 after antithrombotic therapy and recurrence or worsening of stroke, difference in sCLEC-2/D-dimer ratio between non-cardioembolic and cardioembolic AIS or TIA, and correlation between baseline sCLEC-2 and outcome (modified Rankin scale score) after 3 months. sCLEC-2 could be a widely useful biomarker to contribute to the progress of precision medicine in clinical practice of AIS and TIA.

DETAILED DESCRIPTION:
The study design is a multicenter prospective cohort study across Japan including 8 stroke centers. Patients are male or female at age of 20 years or older. The inclusion criteria are (1) AIS within 24 hours of onset and mRS 0 to 2, (2) TIA without MRI positivity within 7 days of onset, and (3) contemporary patients with neurological symptoms, who are required for differentiation from AIS or TIA (served as controls). The main exclusion criteria are (1) platelet or coagulation abnormalities, (2) hemorrhagic stroke, head or other trauma, post-surgery, and hemorrhagic tendency, (3) severe infection, (4) inappropriate patients who were judged by doctors, and (5) poor status of blood samples. The target population is 600 in total (AIS 400, TIA 100 and control 100).

The plasma levels of sCLEC-2 are measured with D-dimer, soluble fibrin, and thrombin-antithrombin complex. sCLEC-2 is determined before starting treatment on admission. The modified Rankin Scale (mRS) and NIH Stroke Scale (NIHSS) are evaluated at registration as baseline data. sCLEC-2 as well as mRS and NIHSS are measured at Day 7 or at discharge. mRS is finally evaluated at 3 months. In the controls, plasma levels of sCLEC-2 and the baseline data are collected at entry.

The sCLEC-2 levels are measured for the difference between patients with AIS or TIA and controls, correlation with severity of stroke, correlation with size of infarct, correlation with Age, Blood pressure, Clinical feature, Diabetes, Duration of symptoms (ABCD2) score in TIA, relationship between treatment effect and worsening or recurrence, difference in the sCLEC-2/D-dimer ratio between cardiogenic and non-cardiogenic etiologies, and difference between TOAST subtypes of ischemic stroke. The study protocol has been approved in each ethical committee at stroke centers.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke within 24 hours of onset and modified Rankin Scale 0 to 2
2. Transient ischemic attack without MRI positivity within 7 days of onset
3. Contemporary patients required for differentiation from ischemic stroke or transient ischemic attack

Exclusion Criteria:

1. Platelet or coagulation abnormalities
2. Hemorrhagic stroke, head or other trauma, post-surgery, and hemorrhagic tendency
3. Severe infection
4. Inappropriate patients who were judged by doctors
5. Poor status of blood samples

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit to the department specialized for stroke
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10-11 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Acute Ischemic Stroke and TIA | On admission before treatment
  The ischemic stroke group and TIA group will be compared with the control group to evaluate whether the sCLEC-2 level contributes to the improvement of the diagnostic accuracy of ischemic stroke and TIA.
Evaluation of Antithrombotic Therapy | On 7+/-1 days after admission
  The post-treatment sCLEC-2 levels in patients with acute ischemic cerebrovascular disorders will be compared between patients without worsening/recurrence (effective treatment group) and those with worsening/recurrence during treatment (ineffective treatment group) to evaluate whether sCLEC-2 measurements contribute to the evaluation of the efficacy of antithrombotic therapy.
Comparison of sCLEC-2 /D-dimer ratio between cardiogenic and non-cardiogenic etiologies | On admission before treatment
  The ischemic stroke group and TIA group will be classified into cardiogenic and non-cardiogenic etiologies based on the TOAST classification to evaluate whether the sCLEC-2/ D-dimer ratio contributes to the accuracy of subtype classification.
Correlation of sCLEC-2 levels on admission with outcome of ischemic stroke and TIA at 3 months | On admission before treatment and 3 months after onset
  The relationships between the sCLEC-2 levels on admission and outcomes at 3 months in the ischemic stroke and TIA groups will be evaluated.

SECONDARY OUTCOMES:
Correlation of sCLEC-2 levels on admission with severity of ischemic stroke or TIA | On admission before treatment
  (1) Correlation with ischemic stroke severity (NIHSS), (2) correlation with size of infarct, (3) correlation with ABCD2 score in TIA will be evaluated.
Difference of sCLEC-2 levels among TOAST subtypes of ischemic stroke | On admission before treatment
  sCLEC-2 levels on admission among subtypes of ischemic stroke will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Katsue Suzuki-Inoue, M.D., Ph.D., Principal Investigator — University of Yamanashi; Shinichiro Uchiyama, M.D., Study Chair — Sanno Medical Center/LSI Medience Co.
Locations (9):
- Japan (9):
  - LSI Medience Co., Katori-shi, Chiba
  - Kyushu Medical Center, Fukuoka, Fukuoka
  - Iwate Medical University, Shiwa-gun, Iwate
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi, Kanagawa
  - Mie Prefectural General Medical Center, Yokkaichi-shi, Mie-ken
  - Showa General Hospital, Kodaira-shi, Tokyo
  - Saiseikai Central Hospital, Minato-ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - University of Yamanashi, Chuo-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Uchiyama S, Suzuki-Inoue K, Wada H, Okada Y, Hirano T, Nagao T, Kinouchi H, Itabashi R, Hoshino H, Oki K, Honma Y, Ito N, Sugimori H, Kawamura M. Soluble C-type lectin-like receptor 2 in stroke (CLECSTRO) study: protocol of a multicentre, prospective cohort of a novel platelet activation marker in acute ischaemic stroke and transient ischaemic attack. BMJ Open. 2023 Sep 18;13(9):e073708. doi: 10.1136/bmjopen-2023-073708. PMID 37723115